CLINICAL TRIAL: NCT03209882
Title: Transcranial Infrared Laser Stimulation (TILS) of Prefrontal Metabolism and Function in Post-traumatic Stress Disorder (PTSD)
Brief Title: Transcranial Infrared Laser Stimulation (TILS) of Prefrontal Cognition in Post-traumatic Stress Disorder (PTSD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB approval terminated
Sponsor: The University of Texas at Arlington (Other)
Collaborators: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Fenghua Tian, PhD, Assistant Professor of Research, The University of Texas at Arlington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2017-0512
Record Dates: First submitted 2017-06-30; First posted 2017-07-06 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-06

CONDITIONS: Post-traumatic Stress Disorder (PTSD)
Keywords: Transcranial infrared laser stimulation (TILS); Near-infrared spectroscopy (NIRS)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- One TILS, one sham, and then five TILS interventions (Experimental): Participants first received a TILS intervention, followed by a sham session one week later. Then, participants received another five weekly TILS interventions.
  Interventions: Device: TILS; Device: sham
- One sham, then six TILS interventions (Experimental): Participants first received a sham session, followed by six weekly TILS sessions.
  Interventions: Device: TILS; Device: sham

INTERVENTIONS:
Device: TILS — Continuous-wave laser of a specific wavelength (1064 nm) was administered to the participants' right forehead for 8 minutes. The laser power was 3.4 Watts.
  Other Names: Low-level laser therapy (LLLT)
Device: sham — The sham session consisted of administering the same laser to the participants' right forehead for totally 8 minutes. However, the laser power was turned to be 0 Watts.

SUMMARY:
This study evaluates the effects of transcranial infrared laser stimulation (TILS) on prefrontal metabolism and hemodynamics in veterans with post-traumatic stress disorder (PTSD). The subjects will receive six TILS interventions and one sham intervention in a course of seven weeks.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is often associated with cognitive impairments. It has been indicated that hypoactivity of the prefrontal cortex plays a major role in the disrupted neural circuitry of mood and cognition.

Transcranial infrared laser stimulation (TILS) is a neural type of photobiomodulation that can elevate neuronal metabolism by exciting cytochrome c oxidase (CCO). Veterans with PTSD will receive prefrontal TILS interventions once-per-week for six weeks. They will also receive an additional sham intervention (laser power = 0) that will be randomly assigned into the first two sessions. Broadband near-infrared spectroscopy (bbNIRS) will be used to directly assess the CCO changes during every TILS/sham session.

Veterans' prefrontal functions will be evaluated with short-term memory tasks before and after each intervention. The prefrontal activities will also be imaged by functional near-infrared spectroscopy (fNIRS) to objectively assess the functional changes due to TILS/sham interventions.

ELIGIBILITY:
Inclusion Criteria:

* War-zone and non-war-zone veterans
* Ages 18-60 years old
* Males and females
* Able to read, speak, and understand English
* Medical records showing prior diagnosis of PTSD (here it refers to the records prior to TILS, which will be assessed and obtained in Visit 1)
* Medical records showing diagnosis of PTSD (here it refers to the CAPS-5 record prior to TILS, which will be assessed and obtained in Visit 1)
* On stable doses of any psychotropic medications for at least 4 weeks

Exclusion Criteria:

* Significant physical disability to perform a computerized memory task
* Past/current significant medical/neurological/mental health disorders known to affect cognitive functioning (e.g., stroke, dementia, schizophrenia, AIDS)
* Presence of moderate/severe TBI, defined as having: alteration of consciousness/mental state >24 hours; posttraumatic amnesia >1 day; loss of consciousness >30 minutes; and/or abnormal structural neuroimaging. We will not exclude veterans with mild TBI, which is found in nearly 50% of veterans with PTSD
* Alcohol abuse/dependence for the past 12- months, as determined by the Rapid Alcohol Problems Screen score >0
* Drug abuse/dependence for the past 12- months, as determined by the Drug Abuse Screening Test-10 score >2
* Severe depression (PHQ-9 total score >19), significant risk of suicide (SBQ-R >6), severe headache (PHQ-15, Item e =2), and/or severe dizziness (PHQ-15, Item g =2)
* Opiate use in the month prior to study entry

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fenghua Tian, PhD, Principal Investigator — University of Texas at Arlington
Locations (1):
- Engineering Research Building (ERB), University of Texas Arlington, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Phenotypic data collected from the subjects and secondary analysis of data (if any) will be deposited at the National Database for Clinical Trials related to Mental Illness (NDCT; http://ndct.nimh.nih.gov/). It will include data collected from the subjects' forehead with optical neuroimaging modalities as well as the subjects' performance scores in three short-term memory tasks. Additional data documentation and de-identified data will be deposited for sharing along with phenotypic data, which includes demographics and PTSD scores.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Six months after completion of the project
Access Criteria: Investigators working under an institution with a Federal Wide Assurance (FWA) and could be used for secondary study purposes in PTSD diagnosis and therapy.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 31 veterans were screened for eligibility between October, 2017 and November, 2018. Ten veterans met the inclusion criteria, among them nine completed the study, and one quit after the initial screening for family reason.
Pre-assignment Details: All of the nine participants were randomly assigned into the two arms.
Period: Overall Study
Arm/Group | One TILS, One Sham, and Then Five TILS Interventions | One Sham, Then Six TILS Interventions
Started | 6 | 3
Completed | 6 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | One TILS, One Sham, and Then Five TILS Interventions | One Sham, Then Six TILS Interventions | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (12.7) | 36.33 (12.7) | 36.3 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 5 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cerebral CCO Changes in Response to TILS and Sham
Description: Cerebral CCO changes measured by broadband NIRS during six TILS interventions and one sham session.
Time Frame: 7 weeks
Measure: Mean (Standard Deviation); unit: microMolar/L
Arm/Group | One TILS, One Sham, and Then Five TILS Interventions | One Sham, Then Six TILS Interventions
Number analyzed (Participants) | 6 | 3
microMolar/L
  Average CCO changes in response to sham | 0.09 (0.21) | -0.33 (0.58)
  Average CCO changes in response to 1st TILS | 0.13 (0.23) | 0.70 (1.22)
  Average CCO changes in response to 2nd TILS | 0.03 (0.27) | 1.44 (2.58)
  Average CCO changes in response to 3rd TILS | 0.04 (0.26) | 2.39 (4.18)
  Average CCO changes in response to 4th TILS | -0.12 (0.57) | 0.86 (1.75)
  Average CCO changes in response to 5th TILS | 0.08 (0.23) | 0.47 (1.01)
  Average CCO changes in response to 6th TILS | 0.09 (0.13) | 1.03 (1.78)

2. Primary Outcome: Cerebral Hemodynamic Changes in Response to TILS and Sham
Description: Cerebral hemodynamic changes measured by broadband NIRS during every TILS or sham session
Time Frame: 7 weeks
Measure: Mean (Standard Deviation); unit: microMolar/L
Arm/Group | One TILS, One Sham, and Then Five TILS Interventions | One Sham, Then Six TILS Interventions
Number analyzed (Participants) | 6 | 3
microMolar/L
  Average deoxy-Hb change in response to sham | 0.40 (0.26) | -0.95 (1.85)
  Average oxy-Hb change in response to sham | 0.28 (1.76) | -1.12 (2.56)
  Average oxy-Hb change in response to 1st TILS | 2.80 (1.71) | 2.77 (5.13)
  Average deoxy-Hb change in response to 1st TILS | 0.08 (0.47) | 1.66 (2.03)
  Average oxy-Hb change in response to 2nd TILS | 3.08 (1.57) | 3.58 (3.97)
  Average deoxy-Hb change in response to 2nd TILS | 0.37 (0.27) | 2.52 (3.53)
  Average oxy-Hb change in response to 3rd TILS | 3.97 (1.44) | 2.60 (2.43)
  Average deoxy-Hb change in response to 3rd TILS | 0.12 (0.21) | 3.37 (5.42)
  Average oxy-Hb change in response to 4th TILS | 2.92 (2.19) | 2.77 (3.01)
  Average deoxy-Hb change in response to 4th TILS | 0.21 (0.48) | 1.89 (3.51)
  Average oxy-Hb change in response to 5th TILS | 2.44 (1.23) | 3.05 (1.45)
  Average deoxy-Hb change in response to 5th TILS | 0.64 (0.54) | 1.04 (2.26)
  Average oxy-Hb change in response to 6th TILS | 2.73 (1.60) | 4.93 (4.10)
  Average deoxy-Hb change in response to 6th TILS | 0.07 (0.65) | 1.31 (3.61)

3. Secondary Outcome: Short-term Memory Scores
Description: The participant's recall time in Digit Forward (DF) task and Digit Backward (DB) task was recorded recorded during initial baseline, and after the one sham and six TILS sessions.
  The recall time indicates how fast the participants could recall that digital numbers 10 seconds after they vanished on computer screen.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: second
Arm/Group | One TILS, One Sham, and Then Five TILS Interventions | One Sham, Then Six TILS Interventions
Number analyzed (Participants) | 6 | 3
second
  DF recall time, baseline | 7.1 (2.9) | 6.5 (3.4)
  DB recall time, baseline | 10.8 (4.8) | 9.5 (3.7)
  DF recall time, sham | 5.4 (1.3) | 5.7 (2.5)
  DB recall time, sham | 8.1 (2.7) | 8.6 (3.3)
  DF recall time, 1st TILS | 6.1 (2.3) | 5.9 (3.3)
  DB recall time, 1st TILS | 8.4 (2.9) | 9.9 (6.9)
  DF recall time, 2nd TILS | 5.6 (1.4) | 5.9 (2.8)
  DB recall time, 2nd TILS | 8.4 (2.7) | 9.2 (5.8)
  DF recall time, 3rd TILS | 5.2 (1.1) | 5.9 (3.5)
  DB recall time, 3rd TILS | 7.4 (1.7) | 11.1 (7.3)
  DF recall time, 4th TILS | 5.0 (1.0) | 6.3 (3.1)
  DB recall time, 4th TILS | 6.3 (1.0) | 7.9 (5.0)
  DF recall time, 5th TILS | 5.1 (0.9) | 5.6 (3.4)
  DB recall time, 5th TILS | 6.2 (1.2) | 8.5 (5.5)
  DF recall time, 6th TILS | 4.9 (0.6) | 5.7 (3.3)
  DB recall time, 6th TILS | 6.5 (1.5) | 7.9 (4.6)

4. Secondary Outcome: Prefrontal Activations in Short-term Memory Processing
Description: Anterior prefrontal hemodynamic activations (HbO2 and Hb changes) measured by functional NIRS during the Digit Forward (DF) and Digit Backward (DB) tasks. The activations were recorded from initial baseline, and after the one sham and six TILS sessions. In post-experiment processing, the activations were averaged in the recall phase, which was a key component related to PTSD.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: microMolar/L
Arm/Group | One TILS, One Sham, and Then Five TILS Interventions | One Sham, Then Six TILS Interventions
Number analyzed (Participants) | 6 | 3
microMolar/L
  DF HbO2, baseline | 0.5 (2.2) | 0.5 (1.4)
  DF Hb, baseline | -0.4 (0.4) | -0.8 (1.5)
  DB HbO2, baseline | 1.4 (2.2) | -0.5 (2.0)
  DB Hb, baseline | 0.7 (1.0) | 0.3 (0.5)
  DF HbO2, sham | -0.6 (3.1) | -2.3 (1.7)
  DF Hb, sham | 0.0 (0.7) | -0.3 (0.4)
  DB HbO2, sham | -1.1 (2.7) | -0.7 (1.1)
  DB Hb, sham | -0.1 (1.2) | 0.2 (0.4)
  DF HbO2, 1st TILS | 0.0 (2.0) | -1.2 (1.3)
  DF Hb, 1st TILS | 0.0 (0.5) | 0.1 (0.5)
  DB HbO2, 1st TILS | -2.5 (4.0) | -1.4 (4.4)
  DB Hb, 1st TILS | -0.5 (1.3) | 0.4 (1.1)
  DF HbO2, 2nd TILS | -2.6 (0.8) | 0.8 (3.8)
  DF Hb, 2nd TILS | -0.1 (0.6) | -1.1 (2.6)
  DB HbO2, 2nd TILS | 1.0 (2.0) | 3.9 (9.6)
  DB Hb, 2nd TILS | 0.7 (1.1) | 2.2 (3.5)
  DF HbO2, 3rd TILS | -1.0 (1.7) | 0.6 (4.0)
  DF Hb, 3rd TILS | -0.2 (0.3) | 0.8 (0.2)
  DB HbO2, 3rd TILS | -3.3 (2.2) | -1.0 (1.0)
  DB Hb, 3rd TILS | -1.1 (1.1) | 0.1 (0.4)
  DF HbO2, 4th TILS | -1.6 (2.8) | -1.8 (1.8)
  DF Hb, 4th TILS | 0.1 (0.7) | 0.1 (0.3)
  DB HbO2, 4th TILS | -1.3 (3.4) | -1.1 (3.7)
  DB Hb, 4th TILS | -0.1 (0.6) | -0.8 (1.0)
  DF HbO2, 5th TILS | -3.2 (2.0) | 0.6 (2.0)
  DF Hb, 5th TILS | -0.3 (1.0) | 0.4 (0.3)
  DB HbO2, 5th TILS | -2.8 (3.5) | 0.6 (3.0)
  DB Hb, 5th TILS | 0.2 (1.0) | 0.4 (0.5)
  DF HbO2, 6th TILS | -2.0 (1.2) | -0.4 (1.5)
  DF Hb, 6th TILS | -0.1 (0.9) | 0.4 (0.7)
  DB HbO2, 6th TILS | 0.4 (2.9) | -5.7 (8.4)
  DB Hb, 6th TILS | 0.2 (1.4) | 0.3 (0.3)

ADVERSE EVENTS:
Time Frame: Entire course of TILS/sham sessions (7 weeks).
Description: The subjects were closely monitored in regard to physical reactions to TILS, and worsening symptoms. A 10-level VAS scale was used to measure headache and dizziness following each TILS/sham session. Severe reaction was defined as VAS ≥5. Then, the subjects were assessed for worsening PTSD symptoms (an increase of ≥24 points in Mississippi-Military), severe depression (PHQ-9 > 19), risk of suicide(SBQ-R ≥ 7).
Arm/Group | One TILS, One Sham, and Then Five TILS Interventions | One Sham, Then Six TILS Interventions
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 0/6 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT03209882/Prot_002.pdf
  • Statistical Analysis Plan (2021-05-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT03209882/SAP_003.pdf